CLINICAL TRIAL: NCT02680145
Title: Prediction of Postsurgical Symptomatic Outcomes With Preoperative Pessary Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John A. Occhino, Assistant Professor of Obstetrics-Gynecology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-006186
Record Dates: First submitted 2016-02-03; First posted 2016-02-11 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Vaginal Vault Prolapse; Pelvic Organ Prolapse; Uterine Prolapse; Pelvic Floor Prolapse
Keywords: Pessary; Prolapse; Cystocele
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse; Prolapse; Cystocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Preoperative Pessary Use (Experimental): All patients will use a pessary for 1-4 weeks preoperatively to reparative surgery for pelvic organ prolapse
  Interventions: Device: Preoperative Pessary Use

INTERVENTIONS:
Device: Preoperative Pessary Use — Pessary use for 1-4 weeks prior to surgical prolapse repair

SUMMARY:
This is a single center, prospective trial of pessary use prior to reconstructive pelvic floor surgery for pelvic organ prolapse. The goal of the study is to evaluate the change in pelvic floor symptoms with pessary use and subsequent reconstructive surgery. Additionally, we will assess the impact that preoperative pessary use has on patient self-reported preparedness for surgery.

DETAILED DESCRIPTION:
It is anticipated that this trial will define the clinical utility of routine preoperative pessary placement, and by shaping patient expectations and increasing preparedness for surgery, we anticipate improving satisfaction and quality of life.

At the initial office visit baseline symptoms are evaluation with validated questionnaire.

The patients' will undergo pessary fitting at least 7 days (but no more than 28 days) prior to scheduled surgical prolapse repair.

Symptomatic change from baseline will be assessed with validated questionnaire preoperatively.

The pessary will be removed at the time of surgery, and the patient will undergo surgical correction of their pelvic organ prolapse (including all restorative surgical procedures, abdominal and transvaginal). A concomitant anti-incontinence procedure will be performed at the discretion of the treating physician in consultation with the patient.

The patients' symptomatic outcome from surgery will then be reassessed by validated questionnaire at 6 weeks and 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* With symptomatic pelvic organ prolapse
* Electing for surgical repair of pelvic organ prolapse (transvaginal or transabdominal) at least 7 days after office consultation
* Understand and have signed written informed consent for preoperative pessary placement.

Exclusion Criteria:

* Previous use of a pessary for pelvic organ prolapse
* Patients undergoing obliterative prolapse surgery (i.e. Colpocleisis),
* Are scheduled for surgery for pelvic organ prolapse less than 7 days after office consultation or greater than 4 weeks after office consultation
* Have an isolated rectocele
* Have allergies to both latex and silicone
* Have an active pelvic infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Occhino, MD, MS, Principal Investigator — Mayo Clinic; Brian Linder, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoperative Pessary Use
Started | 58
Completed | 47
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Preoperative Pessary Use
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 56
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression of Improvement (PGI-I) Score
Description: Number of participants considered treatment success assessed using the 7-point Likert scale of the Patient Global Impression of Improvement (PGI-I) of 1= very much better and 7=very much worse. Patient's will be considered treatment success if they answer "much better" or "very much better" on the PGI-I scale.
Time Frame: 3 months postoperatively
Population: 40 participants completed the PGI-I form 3 months after surgery for data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Pessary Use
Number analyzed (Participants) | 40
Participants | 39

2. Primary Outcome: Prolapse Symptom Severity
Description: Mean value of score on self-reported Pelvic Organ Prolapse Distress Inentory-6 (POPDI-6) questionnaire. Minimum scale score = 0; maximum scale score = 100 and a higher score indicates worse outcome.
Time Frame: Baseline, 3 month post surgery
Population: Data was available for analysis on 36 participants which completed questionnaire at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preoperative Pessary Use
Number analyzed (Participants) | 36
score on a scale
  Baseline score | 48.6 (24.7)
  Follow-up score | 7.3 (14.2)
Statistical Analysis 1: Comparison: Preoperative Pessary Use; Baseline score vs Follow-up score; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Bother of Bladder/Vaginal/Bowel Symptoms
Description: Mean value of score on self-reported Floor Impact Questionnaire-7 (PFIQ-7). Minimum scale score = 0; maximum scale score = 100 and a higher score indicates worse outcome.
Time Frame: Baseline, 3 month post surgery
Population: Data was available for analysis on 40 participants which completed questionnaire at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preoperative Pessary Use
Number analyzed (Participants) | 40
score on a scale
  Baseline score | 72.1 (69.2)
  Follow-up score | 18.8 (49.3)
Statistical Analysis 1: Comparison: Preoperative Pessary Use; Baseline score vs Follow-up score; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Overactive Bladder Symptom Score (OABSS)
Description: Mean value of score on self-reported Overactive Bladder Symptom Score (OABSS) questionnaire. Minimum scale score = 0; maximum scale score = 15 and a higher score indicates worse outcome.
Time Frame: Baseline, 3 month post surgery
Population: Data was available for analysis on 32 participants which completed questionnaire at both time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preoperative Pessary Use
Number analyzed (Participants) | 32
score on a scale
  Baseline score | 12.0 (3.9)
  Follow-up score | 9.6 (2.7)
Statistical Analysis 1: Comparison: Preoperative Pessary Use; Baseline score vs Follow-up score; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject through study participation, duration of approximately 3 months after pelvic surgery.
Arm/Group | Preoperative Pessary Use
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 13/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoperative Pessary Use (N=58)
Urinary Incontinence (Renal and urinary disorders) | 4 (4)
Pelvic Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vaginal dryness with itching (Reproductive system and breast disorders) | 1 (1)
Allergic Reaction on abdomen at surgical site (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vaginal Pain (Reproductive system and breast disorders) | 1 (1)
Vaginal Bleeding Post operative (Reproductive system and breast disorders) | 1 (1)
Hyperkalemia post operative (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia post operative (Hepatobiliary disorders) | 1 (1)
Pelvic floor myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Exacerbated chronic constipation (Gastrointestinal disorders) | 1 (1)
Incidental cystotomy repair (1 cm) (Renal and urinary disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Ureteral vaginal fistula (Reproductive system and breast disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT02680145/Prot_SAP_000.pdf